CLINICAL TRIAL: NCT02344771
Title: Perioperative Endothelial Dysfunction in Patients Undergoing Non-cardiac Surgery
Brief Title: Perioperative Endothelial Dysfunction
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Sarah Victoria Ekeløf Busch, MD, Ph.d. student, Zealand University Hospital
Other Study IDs: SBpoetry
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Myocardial Injury
Keywords: Endothelial dysfunction; General Surgery; Perioperative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Elective colon cancer surgery

SUMMARY:
More than one in 100 otherwise healthy patients undergoing non-cardiac surgery will die within 30 days post-operatively, and of these patients 45% will die from vascular causes such as myocardial infarction. The pathogenesis of perioperative myocardial infarction is complex and to date not fully elucidated. The physiological stress response associated with the surgical procedure is believed to be central in the development of perioperative cardiovascular complications. Surgery initiates systemic inflammation, hypercoagulability and increases the production of catecholamines and cortisol. These drastic systemic changes lead to a state of myocardial oxygen supply-demand mismatch, which added to acute endothelial dysfunction and ruptures of vulnerable plaques, may result in myocardial injury.

The endothelium is a regulator of vascular homeostasis, vascular tone and structure and exerts anticoagulant, antiplatelet and fibrinolytic properties. Endothelial dysfunction is characterized by a decreased vascular bioavailability of nitric oxide probably due to an increased degradation of nitric oxide via its interaction with locally produced reactive oxygen species. No clinical studies have investigated whether peri- and postoperative endothelial dysfunction is associated with an increased risk of perioperative myocardial injury. Endothelial dysfunction may be a key element in the development of perioperative myocardial injury.

The aim of this observational clinical study is to closely examine the endothelial function and its dynamics in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

• Patients scheduled for elective colon cancer surgery

Exclusion Criteria:

* Not capable of giving informed consent after oral and written information
* Previously included in the trial
* Surgery within 7 days of the trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population of patients with colon cancer undergoing elective cancer surgery.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline endothelial function (reactive hyperemia index) at 4 days postoperatively | baseline before operation, 4 hours postoperatively and daily assessments day 1-4 after surgery.
  The reactive hyperemia index is assessed non-invasively by the EndoPat system.

SECONDARY OUTCOMES:
Biomarkers of endothelial function: plasma arginine, plasma asymmetric dimethylarginine and plasma tetrahydrobiopterin | before surgery, 4 hours postoperatively and daily assessments on day 1-4 after surgery
Biomarkers of endothelial glycocalyx degradation (syndecan-1, atrial natriuretic peptide) | before surgery, 4 hours postoperatively and daily assessments on day 1-4 after surgery.
Plasma cardiac troponin I | before surgery and one daily assessment on day 1-4 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Busch, MD, Principal Investigator — Department of Surgery, Koge University Hospital, Denmark
Locations (1):
- Department of Surgery, Roskilde Hospital, Roskilde, Denmark

REFERENCES:
- [Derived] Ekeloef S, Larsen MH, Schou-Pedersen AM, Lykkesfeldt J, Rosenberg J, Gogenur I. Endothelial dysfunction in the early postoperative period after major colon cancer surgery. Br J Anaesth. 2017 Feb;118(2):200-206. doi: 10.1093/bja/aew410. PMID 28100523